CLINICAL TRIAL: NCT02843984
Title: Influence of Vaginal Lactoferrin on Amniotic Fluid Cytokines to Avoid Pregnancy Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Alessandro Trentini, PhD, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRUa1GR-2013-00000220-B
Record Dates: First submitted 2016-07-19; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Pregnancy
Keywords: Amniocentesis
MeSH Terms: interventions — Lactoferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A - untreated (No Intervention): The patients will be not treated with vaginal lactoferrin
- B - 4 hrs treatment (Active Comparator): The patients will be administered with a single dose of 300 mg vaginal lactoferrin 4 hours prior to mid-trimester genetic amniocentesis.
  Interventions: Drug: Lactoferrin
- C - 12 hrs treatment (Active Comparator): The patients will be administered with a single dose of 300 mg vaginal lactoferrin 12 hours prior to mid-trimester genetic amniocentesis.
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Lactoferrin
  Arms: B - 4 hrs treatment; C - 12 hrs treatment

SUMMARY:
Objective: To evaluate the influence of vaginal Lactoferrin administration on amniotic fluid concentration of 47 cytokines, chemokines and growth factors.

DETAILED DESCRIPTION:
60 women undergoing genetic amniocentesis will be enrolled at the Obstetric Unit, University of Ferrara. The selected patients will be randomly assigned to receive 300 mg of vaginal Lactoferrin to obtain 3 groups: A, 20 untreated patients; B and C (20 patients each one) respectively treated 4 and 12 h before amniocentesis. Cytokines, chemokines and growth factors concentrations will be quantified by a magnetic bead Luminex multiplex immunoassays panel technology.

Amniotic fluid samples will be obtained by transabdominal amniocentesis and the sample not required for clinical purposes will be centrifuged to remove particulate material and the supernatants will be aliquoted and stored at -80°C until assay.

ELIGIBILITY:
Inclusion Criteria:

* singleton physiological pregnancy;
* maternal age as the only indication to foetal karyotyping

Exclusion Criteria:

* assumption of drugs interfering with the immune system;
* previous miscarriages;
* pregnancy at risk for maternal or foetal disease;
* lactose intolerance.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Amniotic fluid concentration of mediators involved in inflammation | 1 month after the enrollment of patients will be concluded.
  The investigator will measure the amniotic fluid concentration of 47 mediators (cytokines, chemokines and growth factors) involved in the inflammatory process by Luminex multiplex immunoassays. Controls and Lactoferrin-treated patients will be compared by parametric or non-parametric statistical tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetric Unit, University of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No